CLINICAL TRIAL: NCT03895541
Title: Noninvasive Elastography Evaluation of Myocardial Stiffness in Elderly Patients With Isolated Diastolic Heart Failure: New Diagnostic Tool?
Acronym: ELASTOCARDIO2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-04
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Diseases in Old Age
Keywords: heart failure; myocardial rigidity; new diagnosis; ultrasound imaging
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: stratification
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stratification (Other): All patient will have the same intervention. They will be stratified regarding their degree of heart failure gravity.
  Interventions: Diagnostic Test: SuperSonic image

INTERVENTIONS:
Diagnostic Test: SuperSonic image — 3 examen performed assessed to compared evaluation type: Cardiac magnetic resonance imaging, standard ultrasound imaging and ultrafast imaging

SUMMARY:
The new approach propose in this protocol is based on ultrafast ultrasound and remote palpation of tissue by ultrasonic radiation pressure. Ultrafast ultrasound of biological tissues is based on an innovative ultrasound imaging approach that can image very fast soft tissue events at a rate of several thousands of frames per second and provide quantitative mapping of the elasticity of the tissues. This current project aims is to focus on myocardial rigidity in diastole to better assess the function of the heart failure.

DETAILED DESCRIPTION:
Diastolic heart failure or heart failure with preserved systolic function is the leading cause of heart failure in elderly subjects (more than 2/3 of heart failure in subjects over 60 years). Its main etiology is high blood pressure. Diagnosis of diastolic heart failure remains controversial in clinical practice. It is based on ultrasound and biological criteria. These are mainly acute edema of the lung for patients with preserved Ejection Fraction and high Brain Natriuretic Peptid. It is now recognized that the "primum movens" of this type of heart failure is the increase in myocardial stiffness secondary to left ventricular hypertrophy. The noninvasive evaluation of this parameter would allow a more accurate and reliable diagnosis since it does not depend on the loading conditions, unlike the heart failure and the trans-mitral Doppler). However, the absence of a non-invasive tool for the direct evaluation of diastolic (so-called passive) rigidity prevents the use of this diagnostic parameter. Investigators propose here to non-invasively evaluate the myocardial stiffness in the elderly patient with diastolic heart failure thanks to a new imaging tool using an innovative ultrasonic technology, the ultrafast-echo associated with its elastographic mode "ShearWave Imaging". Investigators have been working for several years in collaboration with the Langevin Institute on this technology, which has recently been validated on experimental models. Its principle is based on the creation of a shear wave from a standard ultrasound probe and the calculation of the velocity of this wave thanks to the very high temporal resolution of the ultrasound system, this speed being correlated to the myocardial rigidity. The human study was recently made possible by the development of a phased array probe with the ability to work with the elastography mode ("ShearWave Imaging").

ELIGIBILITY:
Global Inclusion Criteria:

* Hospitalization in cardiology services for acute pulmonary edema during heart failure
* Natriuretic peptide type B ≥35 pg/ml
* Echocardiographic structural alteration

Specific Inclusion criteria

* Group "preserved LVEF": Left ventricular Ejection Fraction ≥50%
* Group "moderate alteration of LVEF": Left ventricular Ejection Fraction between 40% and 49%
* Group "Systolic heart failure": Left ventricular Ejection Fraction< 40%

Global Exclusion Criteria:

* Other associated lung pathology
* Other heart disease
* Contraindication to MRI or echocardiography gel
* Pregnancy
* Poor echogenicity,

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-01-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Myocardial rigidity assessment | Day 1
  Myocardial rigidity measured using this new non-invasive ultrasound imaging technique.

SECONDARY OUTCOMES:
Norms estimation of myocardial rigidity | Day 1
  Estimation of physiological and pathological norms of myocardial rigidity by elastography
Safety of cardiac elastography | Day 1
  patient monitoring (electrocardiogram scope and constants every10 min) for 30 minutes post-examination associated with a "comfort questionnaire" to be completed by the patient after the examination

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel MESSAS, MD, Principal Investigator — Hopital Européen Georges Pompidou
Locations (1):
- Emmanuel MESSAS, Paris, France

IPD SHARING:
Plan to Share IPD: No